CLINICAL TRIAL: NCT04357093
Title: Evaluation of Remineralizing Efficacy of Grape Seed Extract Oil Versus Fluoride Mouthwash in Management of Post-Orthodontic White Spot Lesions: Randomized Clinical Trial
Brief Title: Remineralizing Efficacy of Grape Seed Extract in Management of White Spot Lesion in Post Orthodontic Treated Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Abd El Sattar Mohamed Kotb, Master degree studnet, Conservative Dentistry Department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Grape seed extract
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape seed extract mouthwash (Experimental): Grape seed extract mouth wash 15% concentration
  Interventions: Other: Grape seed extract mouthwash
- Sodium fluoride mouthwash (Active Comparator): Sodium fluoride mouthwash 1000 ppm
  Interventions: Other: Sodium fluoride mouthwash

INTERVENTIONS:
Other: Grape seed extract mouthwash — Mouthwash 15% grape seed extract
  Other Names: Grape seed extract
  Arms: Grape seed extract mouthwash
Other: Sodium fluoride mouthwash — Sodium fluoride mouthwash
  Arms: Sodium fluoride mouthwash

SUMMARY:
This clinical trial will be conducted to compare the efficacy of grape seed extract oil versus sodium fluoride mouth wash in the management of remineralization in adult patients with white spot lesion over six months.

DETAILED DESCRIPTION:
Natural products have long been used in traditional medicine and are promising sources for novel therapeutic agents, especially in treating oral diseases such as dental caries.

Previously, herbs are used in dentistry for prevention and curative purpose of dental caries. The main advantages of using herbal alternatives are easy availability, cost effectiveness, increased shelf life, low toxicity, and lack of microbial resistance.

Grape seed extract (GSE) has been found to be a promising natural remineralizing agent for treatment of the demineralized tooth.

Grape seed extract (GSE), a readily available over the counter supplement, has been noted for its potential dental restorative and caries preventative properties as a potent antioxidant. There are multiple bioactive properties in GSE, but in particular, its rich content of proanthocyanidins (PACs) plays a role in its theoretical benefit in caries prevention.

PACs have hydrophobic and hydrophilic properties, which enhance their ability to irreversibly bind to a variety of compounds, particularly minerals, proteins, and carbohydrates.

The remineralization effect of GSE appears to be featured. First, it participates in mineral deposition on the superficial layer of the lesion through forming insoluble complexes and combines with calcium to enhance remineralization. Second, GSE may interact with the organic portion of enamel through PA-collagen interaction, thereby stabilizing the exposed collagen matrix.

Proanthocyanidin (PA) has been proved to strengthen collagen-based tissues by increasing collagen cross-links. It is claimed that it can increase collagen synthesis and accelerates the conversion of soluble collagen into insoluble collagen. Proanthocyanidin has proved safe in different clinical applications and has been used as dietary supplements as well.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two WSLs on the labial surfaces of six maxillary anterior teeth that were not present before orthodontic therapy
* Age range between 13 and 30years.

Exclusion Criteria:

* Severe or active periodontal disease.
* Patients had received therapeutic irradiation to the head and neck region.
* Patients had participated in a clinical trial within 6 months before commencement of this trial.
* Patients unable to return for recall appointments
* Presence of abnormal oral, medical, or mental condition.
* Presence of dentin caries or enamel hypoplasia on maxillary anterior teeth.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Remineralization of white spot lesions | Evaluation of tooth surface changes at baseline and at 1, 3 and 6 months after starting treatment .
  changes in fluorescence of white spot lesions will be evaluated after reminerlization by using Diagnodent scoring (0-20)

SECONDARY OUTCOMES:
Satisfaction of the patient: questionnaire | After 6 months
  Using binary questionnaire ( Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt